CLINICAL TRIAL: NCT04241627
Title: Mobile Health Intervention to Promote Medication Adherence Among Adolescents and Young Adults With Chronic Illness
Brief Title: Cell Phone Support to Promote Medication Adherence Among Adolescents and Young Adults With Chronic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Caitlin Sayegh, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-20-00168
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: We will randomly assign participants to cell phone support by voice, cell phone support by text message, or automated text reminders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cell Phone Support (Experimental): An adherence facilitator will deliver Cell Phone Support by daily phone calls Monday through Friday for 12 weeks, to provide social support, medication reminders, problem-solving coaching, incentives for answering calls, and referrals to other services.
  Interventions: Behavioral: Cell Phone Support
- Live Text Support (Experimental): An adherence facilitator will deliver Live Text Support, Monday through Friday for 12 weeks, to provide social support, medication reminders, problem-solving coaching, incentives for answering calls, and referrals to other services.
  Interventions: Behavioral: Cell Phone Support
- Automated Text Reminders (Active Comparator): The comparison condition will include automated text message reminders, using this template: "Take [name of medication] at [set time]. To confirm intake, press REPLY, type CARE 1, and press SEND."
  Interventions: Behavioral: Cell Phone Support

INTERVENTIONS:
Behavioral: Cell Phone Support — Cell Phone Support includes short phone calls (<5 minutes) made each weekday by a human AF to provide social support, medication reminders, problem-solving coaching, incentives for answering calls, and referrals to other services. Cell Phone Support calls focus on assisting AYAs in identifying and accessing resources and support from their natural environments, such as finding ways they can receive needed help from their families, peers, medical teams, and communities. Live Text Support will deliver the same intervention, by text message.
  Other Names: Live Text Support

SUMMARY:
Background: Adolescents and young adults (AYAs) with chronic illnesses often struggle to develop illness self-management skills. Mobile health (mHealth) interventions have been developed for some specific chronic illnesses, but flexible interventions that can be generalized across conditions are needed to accelerate translation.

Research Hypotheses: 1) Cell phone support (CPS) will increase medication adherence and self-management skills across a variety of health conditions; 2) CPS delivered by text message will outperform CPS delivered by phone calls; 3) Patients' perceptions of the human adherence facilitator (AF) will differ based on the mode of communication, text message versus phone calls.

Design: A randomized, controlled, 3-arm pilot trial, following community-based participatory research (CBPR) principles, will test the impact of AF delivered by phone calls or text messages on medication adherence and illness self-management. Conditions will be CPS delivered by phone calls, CPS delivered by text messages, or usual care.

Participants: Participants will include AYAs with diverse chronic illnesses aged 15-20 years (N = 60).

Methods: This study will involve piloting CPS via different communication modes in a randomized trial, informed by CBPR principles. Questionnaires and focus groups will be used to understand how patients perceive the intervention and adherence facilitator.

Main Outcome Measures: Outcomes will include medication and appointment adherence, pharmacy refill ratios, self-management skills, and perceptions of the AF.

Innovation: This study will provide new knowledge regarding how to promote illness self-management skills, and may result in an mHealth intervention with the potential to widely impact supportive care for AYAs with chronic illnesses.

DETAILED DESCRIPTION:
The aim of this randomized pilot trial is to evaluate the acceptability, feasibility, and efficacy of CPS delivered by phone calls or text messages to AYAs with two distinct chronic illnesses, in preparation for an R01 proposal to conduct a multisite, effectiveness-implementation hybrid trial. We propose 1) assessing the feasibility, acceptability, and efficacy of CPS for improving medication adherence, 2) investigating the impact of delivering CPS through live text messages versus phone calls using quantitative and qualitative methods, and 3) evaluating patient and provider views of CPS to guide future implementation work. The proposed research follows the conceptual model, illustrated below, positing that CPS will promote adherence through engaging AYAs in calls or texts with a human AF providing social support. We predict that delivering CPS by text message will increase feasibility and acceptability, perceived social support, and adherence compared to voice delivery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be 1) provider and patient agreement that medication adherence is currently <80%, 2) access to a cell phone, and 3) ability to speak and understand English.

Exclusion Criteria:

* Exclusion criteria will include cognitive impairment that precludes participants from engaging in the consent/assent process or study protocol.

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Sayegh, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Belzer ME, Naar-King S, Olson J, Sarr M, Thornton S, Kahana SY, Gaur AH, Clark LF; Adolescent Medicine Trials Network for HIV/AIDS Interventions. The use of cell phone support for non-adherent HIV-infected youth and young adults: an initial randomized and controlled intervention trial. AIDS Behav. 2014 Apr;18(4):686-96. doi: 10.1007/s10461-013-0661-3. PMID 24271347
- [Result] Sayegh CS, Szmuszkovicz JR, Menteer J, Sherer S, Thomas D, Lestz R, Belzer M. Cell phone support to improve medication adherence among solid organ transplant recipients. Pediatr Transplant. 2018 Jun 19:e13235. doi: 10.1111/petr.13235. Online ahead of print. PMID 29920879
- [Derived] Sayegh CS, MacDonell KK, Iverson E, Beard B, Chang N, Vu MH, Belzer M. Randomized pilot trial of cell phone support to improve medication adherence among adolescents and young adults with chronic health conditions. BMC Digit Health. 2024;2(1):13. doi: 10.1186/s44247-024-00069-w. Epub 2024 Mar 19. PMID 39211575

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cell Phone Support | Live Text Support | Automated Text Reminders
Started | 11 | 12 | 11
Completed | 11 | 12 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cell Phone Support | Live Text Support | Automated Text Reminders | Total
Number analyzed (Participants) | 11 | 12 | 11 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.82 (1.47) | 17.42 (1.62) | 17.82 (1.08) | 17.68 (1.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 16
  Male | 6 | 6 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 6 | 20
  Not Hispanic or Latino | 5 | 4 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 4 | 3 | 3 | 10
  White | 1 | 4 | 0 | 5
  More than one race | 1 | 1 | 4 | 6
  Unknown or Not Reported | 3 | 4 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Medication Adherence
Description: percentage of doses taken out of 100%, reported by the adolescent or young adult, assessed using a visual analogue scale
Time Frame: 12 weeks
Population: Only participants with post-treatment self-report data were analyze for this primary outcome.
Measure: Mean (Standard Deviation); unit: percentage of 100
Arm/Group | Cell Phone Support | Live Text Support | Automated Text Reminders
Number analyzed (Participants) | 11 | 10 | 8
percentage of 100 | 86.55 (17.58) | 84.80 (31.07) | 68.75 (39.03)

2. Primary Outcome: Behavioral Measure of Adherence
Description: percentage of doses taken out of 100%, as measured by the whether participants opened the Medication Event Monitoring System cap the same number of times per day they were prescribed to take medication
Time Frame: 18 weeks
Population: Only participants with who returned their Medication Event Monitoring System cap were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: percentage of 100
Arm/Group | Cell Phone Support | Live Text Support | Automated Text Reminders
Number analyzed (Participants) | 4 | 3 | 3
percentage of 100 | 40.75 (47.14) | 11.67 (12.01) | 14.33 (11.24)

ADVERSE EVENTS:
Time Frame: 1 year post-enrollment in the research study.
Description: We defined adverse event and/or serious adverse event consistently with the clinicaltrials.gov definitions.
Arm/Group | Cell Phone Support | Live Text Support | Automated Text Reminders
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04241627/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04241627/SAP_001.pdf